CLINICAL TRIAL: NCT04299100
Title: Sleep Health Program for Patients With Chronic Pain: A Pilot Randomized Controlled Trial (S-Health)
Brief Title: Sleep Health Program for Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); Unity Health Toronto (Other); Women's College Hospital (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Professor, University of Toronto, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version: Sep 15, 2020
Record Dates: First submitted 2019-11-18; First posted 2020-03-06 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Sleep Disordered Breathing; Chronic Pain; Sleep
MeSH Terms: conditions — Sleep Apnea Syndromes; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants randomized to the Control Group will receive usual care from their pain physician.
- Sleep Health Program - Suspected No/mild sleep apnea (Experimental): Participants randomized to the Sleep Health Program with no/mild sleep apnea.
  Interventions: Behavioral: Sleep Health Program for Participants with No/Mild Sleep Apnea
- Sleep Health Program - Suspected Moderate/severe sleep apnea (Experimental): Participants randomized to the Sleep Health Program with suspected moderate/severe sleep apnea.
  Interventions: Behavioral: Sleep Health Program for Participants with Moderate/Severe Sleep Apnea

INTERVENTIONS:
Behavioral: Sleep Health Program for Participants with No/Mild Sleep Apnea — Participants randomized to the Sleep Health Program will receive the Self-Management for Sleep Care videos and digital materials.
  Other Names: Sleep Health group
  Arms: Sleep Health Program - Suspected No/mild sleep apnea
Behavioral: Sleep Health Program for Participants with Moderate/Severe Sleep Apnea — Participants randomized to the Sleep Health Program with suspected moderate/severe sleep apnea will receive the Self-Management for Sleep Care videos and digital materials, and be recommended for referral to a sleep clinic as part of standard of care.
  Other Names: Sleep Health group
  Arms: Sleep Health Program - Suspected Moderate/severe sleep apnea

SUMMARY:
This is a pilot, prospective, randomized controlled trial of a novel sleep health program versus no sleep intervention in chronic pain patients. The Sleep Health program will consist of weekly home-based videos and digital materials termed "Self-Management for Sleep Care", which will provide participants with information on how to improve their sleep through education on sleep hygiene, relaxation training, and cognitive behavioural components. Patients will be also be screened through undiagnosed sleep apnea. For those determined to have suspected undiagnosed moderate or severe sleep apnea, they will be receive a recommendation for referral to a sleep clinic as part of standard of care. The study aims to evaluate the feasibility and effectiveness of the Sleep Health Program which includes the videos and digital materials and screening for sleep apnea in patients with chronic pain.

DETAILED DESCRIPTION:
All participants will complete sleep, pain, and functional questionnaires. Additionally, all participants will undergo one overnight oximetry reading using the wristwatch pulse oximetry. Following these baseline assessments and questionnaires, participants will be randomized to either the control group or the Sleep Health Program.

A)Sleep Health Program Group Participants in this group will receive usual care from their pain physician. Participants will also receive the Self-Management for Sleep Care videos and digital materials. Participants with suspected moderate/severe sleep apnea as determined by oximetry, but who have not been diagnosed with sleep apnea prior to the study, will be recommended for referral to a sleep clinic as part of standard of care.

B)Control Group Participants in this group will receive usual care from their pain physician.

First follow up visit:

At 8 weeks after the initial visit, all participants will attend their first follow-up visit and complete the sleep, pain and functional questionnaires and 7-day sleep diary recording, and report any changes in medications.

Second follow up visit:

At 6 months after the initial visit, all participants will attend their second follow-up visit and complete the sleep, pain and functional questionnaires, 7-day sleep diary recording and report any changes in medications. Control participants will receive information provided by the Self-Management for Sleep Care program. Control participants with suspected undiagnosed moderate/severe sleep apnea will be recommended for referral to a sleep clinic as part of standard of care.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are:

* Adult patients (≥18 years old) with cognitive capability
* Diagnosed with chronic non-cancer pain for > 3 months
* Reports sleep disturbances such as difficulty falling asleep, staying asleep, or problems waking up too early (responds "Mild", "Moderate", "Severe", or "Very Severe" to items 1, 2, or 3 on the Insomnia Severity Index).

Exclusion Criteria:

* Patients with chronic pain secondary to a neoplasm or metastasis
* Conditions potentially interfering with comprehension and delivery of informed consent, such as certain neurological or psychiatric disorders
* Patients with severe insomnia (Insomnia Severity Index ≥ 22)
* Restless legs syndrome
* Periodic limb movement disorder
* Sleep apnea
* Narcolepsy
* Seizure disorder
* Patients who are pregnant
* Currently undergoing a psychological treatment for insomnia
* Participants who require an urgent sleep physician referral (within four weeks) due to serious medical conditions or safety critical-occupations according to the 2011 Canadian Thoracic Society (CTS) guidelines (e.g. unstable ischemic heart disease, recent cerebrovascular disease, congestive heart failure, refractory systemic hypertension, pulmonary hypertension, hypercapnia respiratory failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of Sleep Health Program | 8 weeks
  Proportion of participants at baseline, and who completed the follow-up visits at 8 weeks.
Feasibility of Sleep Health Program | 6 months
  Proportion of participants at baseline, and who completed the follow-up visits at 6 months.

SECONDARY OUTCOMES:
Efficacy of Sleep Health Program on Functional Outcomes of Sleep Questionnaire-10. | 6 months
  Change from baseline in sleep scores on the Functional Outcomes of Sleep-10 questionnaire at 8 weeks and 6 months. Score range: 0-40, lower score indicates worse functional outcomes.
Efficacy of Sleep Health Program on Insomnia Severity Index | 6 months
  Change from baseline in Insomnia Severity Index score at 8 weeks and 6 months. Score range: 0-28, higher score indicates greater insomnia severity.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, MBBS FRCPC, Principal Investigator — UHN/ University Health Network
Locations (5):
- Canada (5):
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Rehab Institute (TRI), Toronto, Ontario
  - Women's College hospital, Toronto, Ontario
  - Toronto Western Hopsital, Pain Clinic, Dept. of Anesthesia, Toronto, Ontario
  - Mount Sinai Hospital, Department of Anesthesia, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No